CLINICAL TRIAL: NCT04418089
Title: Combination of CAF and Simvastatin Improves Response to Neoadjuvant Chemotherapy and Increases Tumor-Free Margin in Locally Advanced Breast Cancer: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Simvastatin Effect in Combination With Neoadjuvant Chemotherapy to Clinical Response and Tumor-Free Margin in Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Erwin Danil Yulian, Sp.B (K) Onk, Lecturer, Staff of Oncology Division of Department of Surgery, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 18040334
Record Dates: First submitted 2020-05-27; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer; Chemotherapy Effect
Keywords: Simvastatin; Local Advanced Breast Cancer; Clinical Response; Pathological Response; Surgical Margins; Neoadjuvant Chemoterapy
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simvastatin (Experimental): The group received standard treatment with the oral administration of Simvastatin
  Interventions: Drug: Simvastatin 40mg
- Placebo (Experimental): The group received standard treatment with the oral administration of Placebo
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Simvastatin 40mg — The administration of Simvastatin 40 mg in addition to neoadjuvant chemoterapy CAF
  Arms: Simvastatin
Drug: Placebo oral capsule — The administration of Placebo capsule 40 mg in addition to neoadjuvant chemoterapy CAF
  Arms: Placebo

SUMMARY:
Introduction: Neoadjuvant chemotherapy (NACT) has been the standard therapy for treating patients with locally advanced breast cancer (LABC). Doxorubicin-based regimen showed a clinical response for 70-80%. However, the cardiotoxicity from it was not tolerable. Simvastatin acts synergistically with doxorubicin against MCF-7 cells, through downregulation of the cell cycle or induction of apoptosis. Also, it alleviates doxorubicin cardiotoxicity by attenuating ER stress and activating the Akt pathway. Hmgcris a new pathway mediating doxorubicin-induced cell death, and cholesterol control drugs combined with doxorubicin could enhance efficacy and reduce side effects. This study is conducted to see the combination simvastatin and CAF would increase the NACT response and surgical margin of LABC patients.

Methods: This study was a double-blind, randomized placebo-controlled trial, conducted in dr. Cipto Mangunkusumo General Hospital and Koja General Hospital. A total of 70 LABC patients were assessed for eligibility. Patients received either a combination of CAF-Simvastatin (40 mg/day) or CAF-Placebo. The biopsy was taken pre-NACT to make the histopathological diagnosis and examine the expression of HMG-CoA Reductase (Hmgcr) and P-glycoprotein (P-gp). Patients were evaluated for the clinical response after 3 cycles. If the response was positive, patients will proceed to surgery. Then, the post-operative specimen will be reviewed for the pathological response. However, if it was a negative response, patients will be given 2nd line NACT.

DETAILED DESCRIPTION:
Backgrounds Neoadjuvant chemotherapy (NACT) which is followed by surgery is now a standard therapy in the local advanced breast cancer (LABC) since it was introduced 50 years ago, increasingly being used in early-stage LABC patients. Some NACT studies in RSCM use a doxorubicin-based regimen, giving a 70-80% partial response, but do not require a complete response both clinically and pathologically. The NACT response was 80% with a complete clinical response of 36%. The complete pathological response obtained after NACT is the prognosis of a replacement marker both overall and disease-free survival in the LABC. The purpose of giving NACTis to increase tumor resectability and de-escalation surgery and kill micrometastasis which will increase the length of disease-free and life expectancy of the patient. New tumor margins causing post-NACT tumor shrinkage can be used as surgical margins.

Doxorubicin-based chemotherapy is the most commonly given chemotherapy for NACT as well as entering the first line of the National Formulary. However, side effects are limited from drug resistance side effects that can cause cardiomyopathy and heart failure. One of the factors that influence doxorubicin resistance is the presence of efflux pumps such as P-glycoprotein (P-gp) on the cell surface. While the effects of toxicity arise due to the formation of reactive oxygen species (ROS) and the presence of free radicals. Efforts to improve the efficacy of the combination of chemotherapy currently being used with targeted therapies such as anti-HER-2 and bevacizumab, but have a high enough toxicity and are expensive and not included in ForNas. Likewise, some drugs that have been tested in vitro as P-gp inhibitors/modifiers, but failed in clinical trials because of ineffectiveness and greater side effects on the kidneys and heart. Some previous studies have confirmed that simvastatin is a potential ABCB1 / P-gp inhibitor.

Statins are the most widely used anti-hypercholesterolemia in the world, through inhibition of 3-hydroxy-3-methylglutaryl coenzyme-A reductase (Hmgcr) which is an enzyme that limits the use of the mevalonate pathway that can be used as intracellular cholesterol. Besides having pleiotropic effects, statins also have anti-tumor effects. At this time, statins have received approval as a potential anti-tumor agent because several epidemiological studies have agreed on the relationship between statin use and reducing the risk of recurrence of LABC after adjuvant therapy. Some preclinical studies show that statins can decrease breast cancer cell proliferation and induce apoptosis in various experimental models. results from pre-operative "window-of-opportunity" clinical trials on LABC so that statins can reduce tumor proliferation and induce apoptosis. Reports in the RSCM get simvastatin 40 mg for 4 weeks for neoadjuvant reduce the proliferation index in the LABC by 53.3% and inhibit the increase in LABC cells through the Rho / Rock pathway. Although several studios of statin antitumor activity have been carried out, the role of statins in oncology has not yielded satisfactory results or controversies and provides heterogeneous responses depending on the molecular identity and tumor type malignancy. The results of a clinical preliminary study indicate that giving a single statin is not as effective as an anti-cancer because it requires large effects and large side effects.

Several in vitro studies and animal models show that the combination of statins can increase the accumulation of intra-cell chemotherapy so that the effects of potentiation of chemotherapy arise. The administration of a combination of doxorubicin statins increases the potential for anti-cancer effects through the accumulation of doxorubicin in cancer cells, causing the potential for DNA damage, inhibition of proliferation, and induction of apoptosis. statins can also protect cardiotoxic induced by doxorubicin if it is given pre-therapy in mice. With a variety of anti-tumor mechanisms as well as the enormous benefits and potential addition of statins that can be well-tolerated, safe, and inexpensive. However, until now the effects of antiproliferation synergy and induction of apoptosis combination of simvastatin and doxorubicin in LABC patients are not well known. This study aims to determine the efficacy, tolerability, and safety of simvastatin combination and CAF chemotherapy as neo-advanced therapy in LABC patients. The use of this combination is expected to improve clinical and pathological responses as well as surgical margins while providing cardioprotection effects, so as to provide the best service with high oncological value.

Methods

1. Subject and study design This research is a double-blind, placebo-controlled clinical trial conducted at Dr. Cipto Mangunkusumo General Hospital and Koja General Hospital from January 2018 to September 2019. Eligible patients are patients with grade IIIA to IIIC invasive breast cancer that is histologically proven. A total of 60 LABC patients were included in this study. Participants received a combination of NACT CAF and Simvastatin (40 mg / day) (n = 30) or placebo (n = 30). Besides being used to make a histopathological diagnosis, samples were taken by biopsy before NACT, examined for the expression of HMG-CoA Reductase (HMGCR) and P-glycoprotein (P-gp). Participants were evaluated for the clinical response after 3 NACT cycles. If it gives a complete or partial response, then the patient will proceed to surgery. Then, the postoperative specimen will be reviewed for a pathological response. However, if it is stable or progressive, the patient will be given a 2nd line NACT.
2. Tumor assessment The primary outcome was clinical response while the secondary outcome was the pathological response, incision boundary, P-gp expression, Hmgcr expression and side effects. The analysis was performed on the population per protocol. Clinical response assessment uses WHO 1979 criteria. Pathological responses of tumors are evaluated according to the Miller-Payne scoring system. MPG classification is used to evaluate the relevance between pathological response and clinical response. The incision boundary assessment is performed using histopathological tissue incisions depending on the surgical margins of the tumor on the medial, lateral, cranial, caudal, and baseline sides of the tumor; based on the size of the new tumor. Histopathological results will determine whether the level is free from the tumor or not based on the size of the new tumor. Disease assessment is carried out by investigation after 3 NACT cycles. Side effects were assessed during treatment and for 7 days after the last treatment dose and assessed using CTCAE 3.0.
3. Biomarker assessment Estimation of P-glycoprotein (Pgp) and Hmgcr expression was seen under a microscope from a sample after a core biopsy was performed before starting chemotherapy. P-gp expression was interpreted based on the percentage of p-glycoprotein positive cells in the total cell population (low = 0%, 1+ = 1-19%, and 2 + = 20-100% positive cells). Hmgcr expression is interpreted based on the percentage of Hmgcr positive cells in the total cell population (negative = 0%, 1+ = 1-10%, 2+ = 11-50%, 3+ => 51-100% positive cells)..
4. Statistical analysis The main results in this study were clinical responses based on WHO 1970 criteria. ORR values in this study were calculated from the ratio of the number of patients who showed a response (complete and partial) to the total number of patients and were analyzed using the Pearson Chi-Square Test. Secondary outcomes in the form of pathological responses based on GMP and incision boundaries were analyzed using Fisher's Exact Test. Bivariate analysis of clinicopathological variables and molecular biology with the therapeutic response using the Continuity Correction Test and the Fischer's Exact Test. The results of the bivariate analysis with p> 0.25 were performed multivariate analysis using the Logistic Regression Test. The analysis was performed with the help of a computer using the SPSS 23 program. Differences were stated to be meaningful and obtained p values <0.05.

ELIGIBILITY:
Inclusion Criteria:

* LABC IIIA-IIIC TNM / AJCC 2018 with histopathological examination.
* Patients are planned to get NACT
* Performance status of Eastern Cooperative Oncology Group (ECOG) 0-2.
* LABC patients who have not received surgery, radiation or systemic therapy and previous statin therapy.
* Normal kidney organ function (serum creatinine ≤ 1.5 upper limit normal).
* Normal liver organ function (ALT ≤ 2 times the normal limit, or total bilirubin level ≤ 1.5 times the normal upper limit)
* Heart function (E / F)> 55%
* Willing to participate in this study by signing an informed consent

Exclusion Criteria:

* LABC patients are both residual and recurrent.
* Allergy to tattoo ink
* Allergy to statins
* Patients are pregnant or breastfeeding

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-09-05 (Actual)

PRIMARY OUTCOMES:
Clinical Response as WHO 1979 | 3 months
  Clinical Response is measured using WHO 1979 criteria.
  1. Complete Response (CR): Disappearance; confirmed at 3 months
  2. Partial Response (PR): 50% decrease; confirmed at 3 months
  3. Stable Disease(SD): Neither PR nor PD criteria met
  4. Progressive Disease (PD):25% increase; no CR, PR, or SD documented before increased disease

SECONDARY OUTCOMES:
Pathological Response as Measured by Miller-Payne system | 3 months
  Evaluation of the MP system is based on the reduction of tumor cellularity before and after chemotherapy, divided into:
  1. Grade 1 ie there is no change or reduction in cancer cells.
  2. Grade 2: reduction of <30% cancer cells
  3. Grade 3: reduction of cancer cells between 30-90%
  4. Grade 4: reduction of > 90% cancer cells
  5. Grade 5 is that there are no residual cancer cells. Grade 4 is categorized as partial pathology response. Grade 5 is categorized as a complete pathology response
Surgical margin as measured by histopathological | 3 months
  histopathologically the tissue to the tumor incision limit on the medial, lateral, cranial, and caudal sides along with the tumor base; based on the size of the new tumor. Hisopathologically assesses the extent of incision free or not tumor based on the size of the new tumor.
Association of P-gp expression with response by WHO criteria | 3 months
  Clinical Response is measured using WHO 1979 criteria.
  1. Complete Response (CR): Disappearance; confirmed at 3 months
  2. Partial Response (PR): 50% decrease; confirmed at 3 months
  3. Stable Disease(SD): Neither PR nor PD criteria met
  4. Progressive Disease (PD):25% increase; no CR, PR, or SD documented before increased disease
Association of Hmgcr expression with response by WHO criteria | 3 months
  Clinical Response is measured using WHO 1979 criteria.
  1. Complete Response (CR): Disappearance; confirmed at 3 months
  2. Partial Response (PR): 50% decrease; confirmed at 3 months
  3. Stable Disease(SD): Neither PR nor PD criteria met
  4. Progressive Disease (PD):25% increase; no CR, PR, or SD documented before increased disease

CONTACTS AND LOCATIONS:
Overall Officials: Nurjati Chairani Siregar, MD, Study Chair — Department of Pathology, Dr. Cipto Mangunkusumo General Hospital, Jakarta, Indonesia; Baju Adji, Study Chair — Department of Surgery, Koja General Hospital, Jakarta, Indonesia; Filipus Dasawala, MD, Study Chair — Department of Surgery, Dr. Cipto Mangunkusumo General Hospital, Jakarta, Indonesia; Hanifah Hasan, MD, Study Chair — Internship Program as Research Assistant, Department of Surgery, Dr. Cipto Mangunkusumo General Hospital, Jakarta, Indonesia; Muhammad Rizki Kamil, MD, Study Chair — Internship Program as Research Assistant, Department of Surgery, Dr. Cipto Mangunkusumo General Hospital, Jakarta, Indonesia
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No